CLINICAL TRIAL: NCT00169858
Title: Open Randomised Clinical Study of the Long Term Immunogenicity of Engerix-B in 10 Year Old Children and of the Effect of Booster Injections Given 5, 10 or 15 Years After Primary Vaccination
Brief Title: Long Term Immunogenicity Study of Engerix-B Vaccine in 10 Year Old Children and the Effect of Booster Injections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Institut National en Santé Publique du Québec (Other); Centre de Recheche du Centre Hospitalier Université Laval (Other); SmithKlinBeecham Biologicals (Unknown)
Responsible Party: Principal Investigator, Vladimir Gilca, MD, PhD, Laval University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HBV-257 ext. HBV-278; 103860/257 ext. 278
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Hepatitis B; Vaccination
Keywords: Hepatitis B; Vaccination; Engerix-B; Immunogenicity; Long-term immunity; Booster dose; Safety
MeSH Terms: conditions — Hepatitis B | interventions — Engerix-B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Engerix-B — 10 mkg per dose; 3 doses according to 0, 1, 6 month schedule; booster doses 5, 10 or 15 years post-primary vaccination.

SUMMARY:
Hepatitis B immunization has been offered to all grade 4 students (age 9-10) in the province of Quebec, using Engerix-B at a dose of 10 mkg. The peak incidence of hepatitis B occurs between age 15 and 35; the proportion of vaccinated children who will still be protected at this age is currently unknown. This study is designed to determine:

* persistence of immunity until age 25
* persistence of immunological memory as demonstrated by an anamnestic response following a booster dose
* the effect of a booster dose on immunogenicity at either 5, 10 or 15 years after the primary vaccination course (at age (15, 20 or 25).

DETAILED DESCRIPTION:
Three doses of Engerix-B vaccine (10 mkg) were administered according to 0, 1, 6 month schedule to 1126 9-10 year-old children.

The primary objective of the study is to evaluate the persistence of antibodies to Engerix-B in all subjects at age 25 and to compare the levels obtained in those given a booster injection at age 15 or 20 with those receiving no booster injection.

Secondary objectives

* To determine the antibody levels obtained following primary vaccination and the proportion of children who seroconvert
* To determine the antibody levels of one third of subjects at age 15, 5 years after primary vaccination (Group A)
* To determine the effect on antibody levels of a booster injection at age 15 years given to one third of the subjects (Group A)
* To determine the antibody levels of subjects in groups A and B at age 20, 5 years after booster (Group A), 10 years after primary vaccination (Group B)
* To determine the effect on antibody levels of a booster injection at age 20 years given to one third of the subjects (Group B)
* To determine the effect on antibody levels of a booster injection at age 25 years given to one third of the subjects (Group C)
* To determine the antibody levels of subjects in Group A and Group B one year after their 5 or 10 year booster
* To evaluate safety

ELIGIBILITY:
Inclusion Criteria:

* Previously completed the 1995 to 1996 Hepatitis B vaccination program vaccinations (Primary study) to the best of his/her knowledge and already enrolled and followed in the long term study
* Must be HBc negative
* Required standard interval between last dose of primary immunization and booster vaccination
* Written informed consent obtained from the subject
* Free of obvious health problems as established by medical history and clinical examination before entering into the study
* Previously completed routine childhood vaccination to the best of his/her knowledge
* If the subject is female, and the potential of pregnancy exists, it must be asked prior to immunization by the study nurse. According to the protocol d'immunisation du Québec, Engerix-B is not contra-indicated during pregnancy. However, if a participant thinks she could be pregnant (sexually active and no oral contraception or intra uterine device), a pregnancy test will be carried out. In case of pregnancy, the booster vaccination will be performed after delivery.

Exclusion Criteria:

- Not applicable

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1129 (Actual)
Dates: Start 1995-09; Primary Completion 2011-10 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the persistence of antibodies to Engerix-B in all subjects at age 25 and to compare the levels obtained in those given a booster injection at age 15 or 20 with those receiving no booster injection. | 1995 - 2011
  Long term persistence of anti-HBs and the effect of a booster dose given 5, 10 or 15 years post-primary vaccination.

SECONDARY OUTCOMES:
- To determine the antibody levels obtained following primary vaccination and the proportion of children who seroconvert | 1 month post primary vaccination
  Anti-HBs titers were measured 1 months post-primary vaccination
- To determine the antibody levels of one third of subjects at age 15, 5 years after primary vaccination (Group A) | 2001
  Anti-HBs titers were measured 5 years post primary vaccination.
- To determine the effect on antibody levels of a booster injection at age 15 years given to one third of the subjects (Group A) | 2001
  The effect of a booster dose was measured
- To determine the antibody levels of subjects in groups A and B at age 20, 5 years after booster (Group A), 10 years after primary vaccination (Group B) | 2006
  Anti-HBs titers were measured 10 years post primary vaccination (Group B) and 5 years post booster dose (Group A)
- To determine the effect on antibody levels of a booster injection at age 20 years given to one third of the subjects (Group B) | 2006
  Anti-HBs titers were measured 1 month post booster dose given 10 years post-primary vaccination
- To determine the persistence of antibody 15 years after primary vaccination (Group C) | 2011
  Anti-HBs titers will be measured
- To determine the antibody levels of subjects in Group A and Group B one year after their 5 or 10 year booster | 2011
  anti-HBs titers will be measured 10 years post booster dose (Group A) and 5 years post booster dose (Group B)
- To evaluate the effect of a booster dose given 15 years post primary vaccination (Group C) | 2011
  Anti-HBs titers will be measured one month post booster dose (Group C)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Duval, MD, Principal Investigator — Laval University Hospital Center, Public Health Research Unit
Locations (1):
- Vladimir Gilca, Québec, Quebec, Canada

REFERENCES:
- [Result] Duval B, Gilca V, Boulianne N, De Wals P, Masse R, Trudeau G, De Serres G. Comparative long term immunogenicity of two recombinant hepatitis B vaccines and the effect of a booster dose given after five years in a low endemicity country. Pediatr Infect Dis J. 2005 Mar;24(3):213-8. doi: 10.1097/01.inf.0000154329.00361.39. PMID 15750456
- [Result] Duval B, Boulianne N, De Serres G, Laflamme N, De Wals P, Masse R, Trudeau G, Delage G, Desjardins L. Comparative immunogenicity under field conditions of two recombinant hepatitis B vaccines in 8-10-year-old children. Vaccine. 2000 Feb 14;18(15):1467-72. doi: 10.1016/s0264-410x(99)00422-3. PMID 10618544
- [Result] Gilca V, De Serres G, Boulianne N, De Wals P, Murphy D, Trudeau G, Masse R, Duval B. Antibody kinetics among 8-10 years old respondents to hepatitis B vaccination in a low endemic country and the effect of a booster dose given 5 or 10 years later. Vaccine. 2009 Oct 9;27(43):6048-53. doi: 10.1016/j.vaccine.2009.07.100. Epub 2009 Aug 13. PMID 19683086
- [Result] Gilca V, De Serres G, Boulianne N, Murphy D, De Wals P, Ouakki M, Trudeau G, Masse R, Dionne M. Antibody persistence and the effect of a booster dose given 5, 10 or 15 years after vaccinating preadolescents with a recombinant hepatitis B vaccine. Vaccine. 2013 Jan 7;31(3):448-51. doi: 10.1016/j.vaccine.2012.11.037. Epub 2012 Dec 1. PMID 23206974